CLINICAL TRIAL: NCT00840814
Title: Development of a Lymphedema Symptom Checklist in Head and Neck Cancer Patients
Brief Title: Developing a Checklist of Lymphedema Symptoms in Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jie Deng, RN, BSN, MSN, Vanderbilt University
Other Study IDs: CDR0000612406; P30CA068485 (NIH); VU-VICC-SUPP-0834; VU-VICC-080206
Record Dates: First submitted 2009-02-07; First posted 2009-02-10 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Cancer; Lymphedema
Keywords: lymphedema; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
RATIONALE: Developing a symptom checklist for late-effect lymphedema may help doctors learn more about lymphedema in patients with head and neck cancer and plan the best treatment.

PURPOSE: This phase I/II trial is developing a checklist of lymphedema symptoms in patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop and validate a symptom checklist for late-effect lymphedema in patients with head and neck cancer. (Phase I)
* To examine late-effect lymphedema symptoms in these patients using the preliminary patient-symptom checklist developed in phase I. (Phase II)
* To examine the psychometric properties of the patient symptom checklist. (Phase II)

OUTLINE:

* Phase I: Experts review an initial symptom checklist for late-effect lymphedema symptoms and provide suggestions concerning its revision. The checklist is further revised using the card sorting method. Patients sort cards labeled with symptoms into groups that they feel are appropriate based upon their own symptom experiences. Sorting is performed according to frequency and severity of symptoms. Patients may write down any symptoms which are not listed on the cards.

Patients undergo collection of demographic and lymphedema-related symptom information. Additional medical information is obtained from patients' medical records.

* Phase II: A final symptom checklist for late-effect lymphedema symptoms is constructed based on the preliminary checklist developed in phase I. The psychometric properties of the preliminary checklist are also assessed.

Patients undergo collection of demographic, lymphedema-related symptoms, and medical information as in phase I.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patients meeting the following criteria:

    * Diagnosis of local squamous cell carcinoma of head and neck
    * Developed lymphedema after cancer treatment
    * No current evidence of cancer recurrence
    * No metastatic disease
    * Identified from oncology practices at the Vanderbilt-Ingram Cancer Center
  * Volunteer expert meeting the following criteria:

    * Member of the Pain and Symptom Management Team at Vanderbilt-Ingram Cancer Center OR faculty member/clinician associated with the Principal Investigator's prior clinical research at Vanderbilt Medical Center
    * Knowledgeable about the symptoms head and neck cancer patients experience

PATIENT CHARACTERISTICS:

* No history of psychotic illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior cancer treatment
* No concurrent chemotherapy or radiotherapy
* No concurrent anti-psychotic medication

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult head and neck cancer survivors and Head and neck cancer experts
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Late-effect lymphedema symptom checklist | cross-sectional study
Psychometric properties of the patient symptom checklist (Phase II) | cross-sectional study

CONTACTS AND LOCATIONS:
Overall Officials: Jie Deng, RN, BSN, MSN, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee